CLINICAL TRIAL: NCT03656796
Title: Effects of Rhythmic Auditory Cueing With Locomotion Training on Cortical Excitability and Behavior in Patients With Parkinson's Disease
Brief Title: Effects of RAC With Locomotion Training on Cortical Excitability and Behavior in Patients With PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201802068RINC
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-03

CONDITIONS: Parkinson's Disease
Keywords: PD; Auditory cueing; TMS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD with freezing of gait (FOG) (Experimental): Intervention will include treadmill training with auditory cues (AC) and treadmill training without auditory cues (NC).
  Interventions: Other: Treadmill training with auditory cues; Other: Treadmill training without auditory cues
- PD without freezing of gait (FOG) (Experimental): Intervention will include treadmill training with auditory cues (AC) and treadmill training without auditory cues (NC).
  Interventions: Other: Treadmill training with auditory cues; Other: Treadmill training without auditory cues
- Healthy subjects (Control) (Experimental): Intervention will include treadmill training with auditory cues (AC) and treadmill training without auditory cues (NC).
  Interventions: Other: Treadmill training with auditory cues; Other: Treadmill training without auditory cues

INTERVENTIONS:
Other: Treadmill training with auditory cues — Participants should walk on the treadmill according to the rhythmic auditory cues (110% step frequency) for 30 min
  Other Names: AC
Other: Treadmill training without auditory cues — Participants should walk in comfortable speed on the treadmill for 30 min.
  Other Names: NC

SUMMARY:
In this study, 51 subjects include 17 freezers,17 non-freezers and 17 aged-matched healthy subjects will be recruited. We will compare the cortical excitability, gait performance, and stepping-in-place performance before and after intervention of auditory cues combined with gait training. The cortical excitability will be assessed by transcranial magnetic stimulation (TMS). The purpose in this study is to investigate the effects of auditory cues with gait training on cortical excitability and rhythmic movements in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background: Parkinson's disease is a common neurodegenerative disease and movement disorder. Due to the degeneration of basal ganglia, patients with Parkinson's disease also demonstrate internal rhythm dysfunction, thus will lead to difficulty in rhythmic movements such as ambulation. To improve the rhythmic movement problems, auditory cues are often used in clinical setting and have been revealed providing benefits in ambulation and freezing problems for PD subjects. Besides, treadmill training is another common intervention to improve gait performance for PD. However, lack studies investigate the effects of auditory cues with locomotion training on brain neurophysiology and scarcer studies investigate the different effects of auditory cues between the freezers and non-freezers.

Objective: To investigate the effects of auditory-cued training on cortical excitability and motor performances in patients with PD. To investigate whether different effects of auditory cues on cortical excitability and motor performance between the freezers and non-freezers.

Methods: We will recruit 17 freezers, 17 non-freezers and 17 healthy elderly. Each participants will receive the trainings under two conditions in random order. There is one week wash-out period between two-trainings. Two-training are (1) treadmill training with concurrent auditory cues: participants should walk on the treadmill according to the rhythmic auditory cues (110% step frequency) for 30 min. (2) treadmill training without any auditory cues: participants should walk in comfortable speed on the treadmill for 30 min. Assessments consist of cortical excitability through transcranial magnetic stimulation (TMS), stepping-in-place test, and walking test, and they will be done before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 20 y/o
* Diagnosed with idiopathic Parkinson's disease
* No hearing impairment
* Able to walk independently without aid
* MMSE above 24

Exclusion Criteria:

* Other neurological disease
* Orthopedic problems affect gait performance
* Psychological disorder
* Unstable cardiovescular and respiratory status
* Dementia
* Visual disturbance affects gait performance
* Contraindication of transcranial magnetic stimulation: family history of epilepsy; head injury; head surgery or metal implant; pacemaker; syncope or migraine with unknown reasons; pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Transcranial magnetic stimulation (TMS) | 40 min
  TMS will be used to evaluate the cortical excitability. TMS parameters include resting motor threshold (RMT), motor evoke potential (MEPs), cortical silent period (CSP), short intracortical inhibition (SICI) and intracortical facilitation (ICF)

SECONDARY OUTCOMES:
10 meter walking test | 10 min
  The foot sensors is used to measure the coefficient of variance of step time (step time CV), gait velocity, stride length, and cadence.
Stepping-in-place test | 5 min
  The foot sensors are used to measure the stepping variability between each step.

CONTACTS AND LOCATIONS:
Overall Officials: Jer-Junn Luh, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhong Cheng, Taiwan